CLINICAL TRIAL: NCT03692169
Title: The Changes of Retinal and Choroidal Capillaries After Half-dose Photodynamic Therapy Measured by Angio- OCT in Eyes With Central Serous Chorioretinopathy
Brief Title: The Changes of Retinal Capillaries After Half-dose PDT Measured by OCTA in Eyes With CSC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jin Chen-jin (Other)
Responsible Party: Sponsor-Investigator, Jin Chen-jin, Jin Chen-jin, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: CSC-PDT-OCTA（ZOC）
Record Dates: First submitted 2018-09-26; First posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Central Serous Chorioretinopathy
Keywords: Central serous chorioretinopathy
MeSH Terms: conditions — Central Serous Chorioretinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- CSC patients: Half-dose photodynamic therapy was performed when a serous retinal detachment involving the macular fovea was present; The treatment field size was set as 3000 microns. This was achieved by administering 3mg/m² of Verteporfin intravenously over a period of 10 minutes. Fifteen minutes after commencing the verteporfin infusion the GLD was exposed to a 689 nm laser light with a florescence of 600 mw/cm² for 83 seconds and a total energy of 50 J/cm². OCTA (XR Optovue, Fremont, CA, USA) and spectral domain OCT (SD-OCT) were performed at baseline and each follow-up (one month and three months) visit after hd-PDT.
  Interventions: Procedure: Half-dose photodynamic therapy

INTERVENTIONS:
Procedure: Half-dose photodynamic therapy — Half-dose photodynamic therapy was achieved by administering 3mg/m² of Verteporfin (Visudyne; Novartis, Switzerland) intravenously over a period of 10 minutes. Fifteen minutes after commencing the verteporfin infusion the greatest linear dimension was exposed to a 689 nm laser light with a florescence of 600 mw/cm² for 83 seconds and a total energy of 50 J/cm². Optical coherence tomography angiography (OCTA) with the split-spectrum amplitude-decorrelation angiography algorithm (XR Optovue, Fremont, CA, USA) and spectral domain OCT (SD-OCT) were performed at baseline and each follow-up (one month and three months) visit after hd-PDT.

SUMMARY:
To determine changes in retinal and choroidal capillaries with optical coherence tomographic angiography (OCTA) after half-dose photodynamic therapy (hd-PDT) in eyes with central serous chorioretinopathy (CSC).

DETAILED DESCRIPTION:
PDT was hypothesized to have a primary effect on the choroidal capillaries, and a number of studies have reported choriocapillary damage and choroidal vascular remodeling after PDT. More recently, although OCTA related CSC research has been conducted, no quantitative report has thoroughly investigated the microstructural changes in the superficial, deep retinal and choroidal capillaries after hd-PDT. The purpose of the present study is to determine the changes in the retinal and choroidal capillaries quantitatively with OCTA after hd-PDT in eyes with CSC.

This is a prospective observational study of patients undergoing hd-PDT for CSC with active leakage in retinal pigment epithelium (RPE) and followed for 3 months. Fundus fluorescein angiography (FFA) and indocyanine green angiography (ICGA) were performed at baseline; best corrected visual acuity (BCVA), fundus photography, optical coherence tomography angiography (OCTA) with the split-spectrum amplitude-decorrelation angiography algorithm (XR Optovue, Fremont, CA, USA) and spectral domain OCT (SD-OCT) were performed at baseline and each follow-up visit after hd-PDT.

ELIGIBILITY:
Inclusion Criteria:

1. CSC diagnosed by FFA and ICGA, where the active leakage was just located in macular fovea with SRF confirmed by OCT
2. Patient age ≥18 years
3. BCVA ≥35 letters on ETDRS charts
4. Persistent CSC for a period of time or patients were anxiety about the symptom and asking for treatment
5. Lack of either spontaneous improvement or improvement induced by empirical treatment such as pharmaceutical drug
6. The provision of written informed consent -

Exclusion Criteria:

1. The presence of any other chorioretinal diseases that may affect the studies, such as age-related macular degeneration (AMD), polypoidal choroidal vasculopathy (PCV)
2. Patients who had received any previous treatment, including PDT, intraocular drug injection or focal thermal laser photocoagulation for CSC
3. Patients with PED in macular fovea which the average diameter (transverse diameter and vertical diameter) was more than 300 microns
4. Patients with high myopia, defined as a refractive error (spherical equivalent) < -6.00 diopters, or an axial length >26.5 mm
5. Patients with media opacities, or signal strength index of the images < 60
6. Patients under corticosteroid therapy -

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Central Serous Chorioretinopathy (CSC)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-10-31 (Actual); Primary Completion 2018-10-10 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes of retinal capillaries after hd-PDT | 1 month, 3 month
  The primary outcome measure is the OCTA-based changes in the retinal capillaries after hd-PDT

SECONDARY OUTCOMES:
The proportion of eyes with complete absorption of subretinal fluid(SRF) | 1 month, 3 month
  The outcome 2 measure is the OCT-based improvement rate (defined as the proportion of eyes with complete absorption of subretinal fluid on OCT images)
Change of Best Corrected Visual Acuity(BCVA) | 1 month, 3 month
  The outcome 3 measure is the EDTRS charts-based improvement of Best Corrected Visual Acuity
Changes of choroidal thickness after hd-PDT | 1 month, 3 month
  The outcome 4 measure is the OCT-based thinning of choroidal thickness after hd-PDT

CONTACTS AND LOCATIONS:
Overall Officials: Chenjin Jin, Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (2):
- China (2):
  - Fabao Xu, Guangzhou, Guangdong
  - Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Peng J, Zhong L, Ma L, Jin J, Zheng Y, Jin C. Comparison of vascular parameters between normal cynomolgus macaques and healthy humans by optical coherence tomography angiography. BMC Ophthalmol. 2019 Oct 11;19(1):204. doi: 10.1186/s12886-019-1207-x. PMID 31601186